CLINICAL TRIAL: NCT03809546
Title: Differential Female Response to Δ9-tetrahydrocannabinol (THC): The Influence of Estradiol
Brief Title: Individual Differences in Drug Response
Acronym: IDT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB18-1286
Record Dates: First submitted 2019-01-11; First posted 2019-01-18 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-01

CONDITIONS: Differential Female Response to Δ9-tetrahydrocannabinol (THC)
MeSH Terms: interventions — Dronabinol; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: dextrose
- 7.5 mg THC (Active Comparator)
  Interventions: Drug: Dronabinol
- 15 mg THC (Active Comparator)
  Interventions: Drug: Dronabinol

INTERVENTIONS:
Drug: Dronabinol — THC (Marinol® [dronabinol]; Solvay Pharmaceuticals) will be orally administered in doses of 7.5 mg and 15 mg, in opaque capsules with dextrose filler. Placebo capsules contain only dextrose. These doses of THC are known to produce performance impairments as well as subjective intoxication with little to no adverse reactions in experienced occasional, but non-daily cannabis users (Ménétrey et al., 2005; Issa et al. 2016).
  Arms: 15 mg THC; 7.5 mg THC
Drug: dextrose — We are administering dextrose to health volunteers for our placebo group
  Arms: Placebo

SUMMARY:
Females are increasingly using cannabis, yet remain underrepresented in preclinical and clinical cannabinoid research. This female-specific research plan will test the effects of two recreationally relevant doses of oral THC and placebo in healthy females at two phases of the menstrual cycle. Acute oral THC will be administered in a double-blind and counterbalanced design. Menstrual cycle phase will be determined using blood serum analyses of estradiol and progesterone and self-reported responses. The main hypothesis is circulating estradiol levels are associated with cardiac, neuroendocrine, and subjective THC response. The rationale for the presented work is to better understand the risks of cannabis use, in order to maximize possible medical potential and minimize public health risks. The expected outcome of this work is a deeper understanding of how circulating estradiol levels may associate with response to THC and how the physiological response is associated with the subjective response. Uncovering the individual differences in response to THC will allow for more preventive action against cannabis-induced anxiety, paranoia, and psychosis.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old, females (N=60)
* Body Mass Index 19-26
* High school education, fluent in English
* Occasional cannabis users ( <11 times in past 30 days)

Exclusion Criteria:

* History of daily cannabis use
* Past or present severe substance use disorder
* Current or past diagnosis with drug treatment for psychosis/bipolar/schizophrenia
* Past year major depression
* Current or past Post Traumatic Stress Disorder
* Attention Deficit Hyperactivity Disorder
* Cardiovascular illness, high blood pressure, abnormal electrocardiagram
* Current medications (NO hormonal birth control or intrauterine device)
* Pregnant or planning to become pregnant

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Pabon, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | 7.5 mg THC | 15 mg THC
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 7.5 mg THC | 15 mg THC | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 60
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 20 | 60
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 3 | 9
  White | 14 | 14 | 14 | 42
  More than one race | 3 | 3 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60
High School Education [Count of Participants; unit: Participants] | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Profile of Mood States (POMS)
Description: The POMS measures individuals' mood states. This is a validated scale to measure positive and negative mood states. The POMS contains 30 items and assess six identified mood factors: Tension-Anxiety, Depression-Ejection, Anger - Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment. Scoring of this instrument provides a global score of 0 to 120 or individual domain scores. Subscale scores range from 0-20. Lower scores indicate better mood state. The POMS brief form is a simple self-rating instrument.
Time Frame: Difference from baseline (time 0 or pre-capsule) to post-capsule (120 min)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 7.5 mg THC | 15 mg THC
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Tension - Anxiety | 2.58 (0.047) | 4.28 (0.07) | 8.25 (0.05)
  Depression - Ejection | 0.7 (0.005) | 1.2 (0.02) | 1.04 (0.004)
  Anger - Hostility | 1.2 (.01) | 1.5 (.025) | 4.25 (.036)
  Vigor - Activity | 5.02 (0.04) | 7.5 (0.05) | 6.25 (0.09)
  Fatigue - Inertia | 2.0 (0.11) | 3.75 (0.04) | 7.25 (0.01)
  Confusion - Bewilderment | 2.0 (0.065) | 2.25 (0.055) | 3.25 (0.04)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 8 weeks
Arm/Group | Placebo | 7.5 mg THC | 15 mg THC
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT03809546/Prot_SAP_000.pdf